CLINICAL TRIAL: NCT00459485
Title: Effects of Initiation and Discontinuation of Short Term Zinc Supplementation on the Magnitude and Velocity of Change in Plasma Zinc Concentration
Brief Title: Effects of Initiation and Discontinuation of Short Term Zinc Supplementation on Plasma Zinc Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Kenneth Brown, University of California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200714985; SerumZinc
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Zinc Deficiency
Keywords: Plasm zinc concentration; Zinc supplementation; Assessment of zinc status; Plasma zinc concentration
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zinc supplement (20 mg) (Experimental): Daily intake of 20 mg supplementary zinc
  Interventions: Dietary Supplement: zinc sulfate
- Zinc supplement (10 mg) (Experimental): Daily intake of 10 mg supplementary zinc
  Interventions: Dietary Supplement: zinc sulfate
- Placebo supplement (Placebo Comparator): Daily intake of placebo supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: zinc sulfate — 20 or 10 mg zinc per day for 3 weeks
  Other Names: Producer: UCD pharmacy
  Arms: Zinc supplement (10 mg); Zinc supplement (20 mg)
Dietary Supplement: Placebo — Daily placebo for 3 weeks
  Other Names: Producer: UCD pharmacy
  Arms: Placebo supplement

SUMMARY:
This is a double-blind, randomized controlled trial conducted in men 19-65 years of age who will receive daily zinc supplements (10 or 20 mg zinc/d as zinc sulfate) or placebo for 21 days. Blood samples for plasma zinc and CRP concentrations will be drawn at baseline and days 1, 2, 5, 9, 14, and 21 during supplementation and days 1, 2, 5, 9, and 14 after discontinuation of supplementation.

DETAILED DESCRIPTION:
The study will be a double blind, randomized, placebo controlled trial conducted in men 19-65 years of age. Participants will receive daily zinc or placebo liquid supplements for 21 days. Supplemental zinc will be given as zinc sulfate; the lower dose zinc supplement will contain 10 mg/d elemental zinc, and the higher dose zinc supplement will contain 20 mg/d elemental zinc. The placebo will contain the same excipients expect for zinc sulfate.

Multiple blood draws will be performed throughout the course of the study, to determine the responsiveness of plasma zinc concentrations to zinc supplementation. Two baseline blood draws will occur prior to the start of supplementation (study days -7 and 0). Blood draws will be performed on days 1, 2, 5, 9, 14 and 21 of the 21 day supplementation period. Upon termination of supplementation (day 21), blood draws will be performed on days 1, 2, 5, 9, 14 and 21 post-supplementation (study days 22, 23, 26, 30, 35 and 42).

The major outcomes of interest are the magnitude and velocity of change in plasma zinc concentration. Other outcomes to be assessed are plasma concentrations of the acute phase proteins CRP and AGP, as well as reported morbidity, because of their potential roles as confounding variables. Anthropometric variables will be assessed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Generally health men
* 19-65 years
* Non-anemic

Exclusion Criteria:

* Age <19 or >65
* Hemoglobin <120 g/L
* Clinical evidence of illness
* Consumption of mineral supplements
* Recent blood donation (within 8 weeks)

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plasma zinc concentration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis

REFERENCES:
- [Derived] Wessells KR, Jorgensen JM, Hess SY, Woodhouse LR, Peerson JM, Brown KH. Plasma zinc concentration responds rapidly to the initiation and discontinuation of short-term zinc supplementation in healthy men. J Nutr. 2010 Dec;140(12):2128-33. doi: 10.3945/jn.110.122812. Epub 2010 Oct 13. PMID 20943956